CLINICAL TRIAL: NCT04310917
Title: Clinico-biological Collection of Subjects With Hyper Lipoprotein a in Reunion Island
Acronym: COLLIPAR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020/CHU/01
Record Dates: First submitted 2020-03-13; First posted 2020-03-17 (Actual); Last update posted 2022-08-30 (Actual); Status verified 2022-08

CONDITIONS: Cardiovascular Disease
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lipoprotein a level (Other): blood lipoprotein (a) test
  Interventions: Other: blood lipoprotein (a) test

INTERVENTIONS:
Other: blood lipoprotein (a) test — research specific blood sample

SUMMARY:
Cardiovascular disease (CVD) is the second leading cause of death in France and the leading cause of death on Reunion Island. Some modifiable risk factors for cardiovascular diseases are well identified and can be easily modulated, in particular by hygiene and dietetic measures (tobacco, sedentary lifestyle). Other risk factors such as high blood pressure, diabetes or dyslipidemia can also be pharmacologically modulated. On the other hand, there is a cardiovascular risk factor that we do not know how to modulate: a high level of lipoprotein (a) (Lp (a)), whose regulation remains largely unknown.

High plasma levels of Lipoprotein (a) remain a major risk for the development of cardiovascular disease and its clinical complications, which no drug can currently reduce. Understanding the biological and genetic determinants modulating Lp (a) levels remains a major challenge for treating subjects with hyper Lp (a). Several individuals and possibly Reunion families have been detected as having abnormally high rates of apo (a)

Thanks to the link between cardiovascular clinical picture, Lp (a) concentration and other biological markers, the study should allow a better understanding of the mechanisms underlying the cardiovascular risk in order to offer advice. prevention and care of at-risk subjects screened; or even avenues for adapted genetic counseling (DNA sequencing).

At the genetic level, several hypotheses could be explored making it possible to link the expression of the apo (a) protein to the genotype, in particular the presence of mutations in the gene, in the promoter region, polymorphisms, or epistatic regulation.

ELIGIBILITY:
Inclusion Criteria:

* Patient with Lp (a)> 200 nmol / L OR member of family of a patient with Lp (a)> 200 nmol / L
* be affiliated or beneficiary of a social security scheme
* signed consent

Exclusion Criteria:

* Refusal to participate

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-09-19 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Carry out a family screening of the plasma Lp (a) level | at inclusion
  Carry out a family screening of the plasma Lp (a) level around index cases followed or directed towards Reunion University Hospital (index case = Lp (a) rate> 200nmol / L)

CONTACTS AND LOCATIONS:
Overall Officials: Ilya KHANTALIN, PH, Principal Investigator — CHU de la Réunion
Locations (1):
- Centre Hospitalier Universitaire de la Réunion, Saint-Denis, France

IPD SHARING:
Plan to Share IPD: No